CLINICAL TRIAL: NCT01522014
Title: Five-Year Outcome of Ceramic on Ceramic Bearing Versus Ceramic on Crossfire® Highly Cross-Linked Polyethylene Bearing in Primary Total Hip Arthroplasty: A Randomized Trial
Brief Title: Randomized Clinical Trial of Ceramic Bearing Primary Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Stryker Canada LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00000886
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Total Hip Replacement
Keywords: Joint Replacement; Health Related Quality of Life; Functional Outcomes; Revision Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceramic on Ceramic (Active Comparator): Subjects received a ceramic on ceramic bearing total hip replacement.
  Interventions: Device: Secure-Fit™ arc-deposited Hydroxylapatite (HA) shell - surface ceramic and an Alumina Bearing Couple (ABC) ceramic insert and Ceramic C-taper head
- Ceramic-on-Highly Crosslinked Polyethylene (Active Comparator)
  Interventions: Device: Secure-Fit™ arc-deposited hydroxylapatite shell, a Crossfire® insert and a Ceramic C-taper head

INTERVENTIONS:
Device: Secure-Fit™ arc-deposited Hydroxylapatite (HA) shell - surface ceramic and an Alumina Bearing Couple (ABC) ceramic insert and Ceramic C-taper head
  Arms: Ceramic on Ceramic
Device: Secure-Fit™ arc-deposited hydroxylapatite shell, a Crossfire® insert and a Ceramic C-taper head
  Arms: Ceramic-on-Highly Crosslinked Polyethylene

SUMMARY:
Primary total hip arthroplasty (THA) has been a very successful surgical intervention in the geriatric population. Numerous studies have reported good mid and long term results of THA in patients over the age of 60 years. With the reported high success rate of this surgical intervention, the THA surgery is being performed in younger patients who have significant joint disease.

A clinical trial, using a randomized blinded design, was undertaken to compare the functional outcome of 1) alumina heads/alumina liners, and 2) alumina head/Crossfire polyethylene liners in patients 60 years of age or younger with non-inflammatory arthritis of the hip.

Subjects were assessed preoperatively and at one and five years postoperatively. Ten-year follow-up is currently underway.

The primary outcome measure is the WOMAC Osteoarthritis Index. Secondary measures were the RAND-12, as well as measurement of complication and revision rates. The patient's demand on the implant as calculated by the patient's age, weight, health status and activity level was also measured.

ELIGIBILITY:
Inclusion Criteria:

* Males or females scheduled for primary THA to treat non-inflammatory arthritis
* Less than 61 years old at time of surgery
* Able to speak and read the English language or have an available translator
* Dorr Index A or B bone quality on preoperative radiographs
* Willing and able to return for follow-up visits

Exclusion Criteria:

* Have femoral or acetabular bone deficiency requiring augmentation
* Ongoing corticosteroid use
* Dorr Index C bone quality on the preoperative radiograph
* Required a prosthesis neck length of greater than five millimeters

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 1997-11; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMaster Osteoarthritis Index (WOMAC) Pain Score | Five Years
  This is a disease-specific, patient reported outcome measure of pain.
WOMAC Function Score | Five years
  This is a disease-specific patient reported outcome measure of function
WOMAC Stiffness Score | Five Years
  This is a disease-specific, patient-reported outcome measure of stiffness.

SECONDARY OUTCOMES:
WOMAC Pain Score | One Year
  This is a disease-specific, patient-reported outcome measure of pain.
WOMAC Function Score | One Year
  This is a disease-specific, patient-reported outcome measure of function.
WOMAC Stiffness Score | One Year
  This is a disease-specific, patient-reported outcome measure of stiffness.
RAND 12-Item Health Survey (RAND-12) | Five Years
  This is a generic patient-reported outcome measure of health status.
RAND-12 | One years
  This is a generic patient-reported outcome measure of health status.
Complications | Five Years
  This measured the postoperative complications.
Revisions | Five Years
  This measured the number of revisions in five years
WOMAC Pain Score | 10 Years
WOMAC Function Scores | 10 years
WOMAC Stiffness Score | 10 years
RAND-12 | 10 years
Complications | 10 years
Revision Rate | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Beaupre, PT, PhD, Study Director — University of Alberta; D William C Johnston, MD, FRCS (C), Principal Investigator — Alberta Health services
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta